CLINICAL TRIAL: NCT02236091
Title: Monitoring Everyday Life Motor Activity in Children
Acronym: MELMAC
Status: Terminated | Type: Observational
Why Stopped: Lacking algorithms led to abortion of project
Sponsor: Rob Labruyere (Other)
Responsible Party: Sponsor-Investigator, Rob Labruyere, PhD, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: MELMAC
Record Dates: First submitted 2014-09-01; First posted 2014-09-10 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Neurologic Disorders
Keywords: cerebral palsy; stroke; traumatic brain injury
MeSH Terms: conditions — Nervous System Diseases; Cerebral Palsy; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inpatients

SUMMARY:
The overall aim of this project is to monitor everyday life activity of children with neurological disorders undergoing rehabilitation using wearable sensors capable of accurate and unobtrusive long-term measurement.

Specific objectives:

1. To adapt the sensors for the use by children with neurological disorders. The focus lies on the exact positioning and the investigation of the needed amount of IMUs.
2. To validate the sensor data with collected video recordings and to develop specific algorithms to automatically extract specific movements and to analyze long-term sensor recordings.
3. To perform a cross-sectional study to assess intensity, task-specificity and duration of upper and lower limb activity during rehabilitation. There, we aim to gain objective information about levels and types of activity during rehabilitation in relation to age, gender and disorder.
4. To conduct a responsiveness study to assess whether or not the sensor output is able to highlight changes over time during rehabilitation.

Therefore, at time point T=0 (shortly after admission to our center), participants are equipped with 3 inertial measurement units (1 at each wrist and 1 at the sternum). Additionally, a small wearable camera is mounted to the chest. The participants then return to their everyday life for 4 hours (no therapies, measurement period is in the evening). Afterwards, the equipment is removed again. To investigate responsiveness, the same protocol is being repeated 4 weeks later (time point T=1).

ELIGIBILITY:
Inclusion Criteria:

* Various neuro-orthopedic diagnoses. Broad inclusion criteria are required to better generalize study results to the patient population of our center.
* Both walking or in wheelchair, but mobility independent from assisting people
* Cognitive ability to be able to follow simple verbal instructions.
* Signed informed consent from legal guardians and also from adolescents aged 15 years or older before study onset.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be inpatients from our rehabilitation center and will be recruited directly by researchers working on this project
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Counts per minute at time point T=0 | At T=0
  From the wearable sensors at the wrist, a count/minute statistic is calculated that reflects the amount of activity the child performs during that time.
Counts per minute at time point T=1 | At T=1 (4 weeks after T=0)
  From the wearable sensors at the wrist, a count/minute statistic is calculated that reflects the amount of activity the child performs during that time.

SECONDARY OUTCOMES:
Motor assessment: Melbourne 2 at time point T=0 | At T=0
  The Melbourne Assessment 2: a test of unilateral upper limb function is a validated and reliable tool for evaluating quality of upper limb movement in children with neurological conditions aged 2.5 to 15 years. For ease of use the assessment's full title is simplified to The Melbourne Assessment 2 or MA2.
  The MA2 is a criterion-referenced test that extends and refines the scale properties of the original Melbourne Assessment. The MA2 measures four elements of upper limb movement quality: movement range, accuracy, dexterity and fluency. It comprises 14 test items of reaching to, grasping, releasing and manipulating simple objects. Each child's test performance is videorecorded for subsequent scoring.
Parent questionnaire: Abilhand-Kids at time point T=0 | At T=0
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved.
Motor assessment: Melbourne 2 at time point T=1 | At T=1 (4 weeks after T=0)
  The Melbourne Assessment 2: a test of unilateral upper limb function is a validated and reliable tool for evaluating quality of upper limb movement in children with neurological conditions aged 2.5 to 15 years. For ease of use the assessment's full title is simplified to The Melbourne Assessment 2 or MA2.
  The MA2 is a criterion-referenced test that extends and refines the scale properties of the original Melbourne Assessment. The MA2 measures four elements of upper limb movement quality: movement range, accuracy, dexterity and fluency. It comprises 14 test items of reaching to, grasping, releasing and manipulating simple objects. Each child's test performance is videorecorded for subsequent scoring.
Parent questionnaire: Abilhand-Kids at time point T=1 | At T=1 (4 weeks after T=0)
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Labruyère, PhD, Principal Investigator — Children's University Hospital Zurich
Locations (1):
- Rehabilitation Center of the Children's University Hospital, Affoltern am Albis, Switzerland

REFERENCES:
- [Background] Strohrmann C, Labruyere R, Gerber CN, van Hedel HJ, Arnrich B, Troster G. Monitoring motor capacity changes of children during rehabilitation using body-worn sensors. J Neuroeng Rehabil. 2013 Jul 30;10:83. doi: 10.1186/1743-0003-10-83. PMID 23899401